CLINICAL TRIAL: NCT02693587
Title: Misodel or Angusta for Induction of Labour? - a Medical Health Technology Assessment
Brief Title: Misodel or Angusta for Induction of Labour?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Holbaek Sygehus (Other)
Collaborators: Naestved Hospital (Other); Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 50213
Record Dates: First submitted 2015-11-09; First posted 2016-02-26 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Safety; Efficacy; Cost; Experience

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Misodel group in Holbæk: Misodel for induction of labour in Holbæk
  Interventions: Drug: Misodel and Angusta
- Angusta group in Roskilde and Næstved: Angusta for induction of labour in Roskilde and Næstved
  Interventions: Drug: Misodel and Angusta

INTERVENTIONS:
Drug: Misodel and Angusta

SUMMARY:
In Denmark, every 4 birth induced, most often due to prolonged pregnancy, up til 10-12 days after term. A group (RADS) set up by the Danish Regions has recently recommended induction with prostaglandins in tablet form (Angusta®). The recommendation is based primarily on the results of a meta-analysis published by the Cochrane Library, where various prostaglandin medications were compared.

Vaginal prostaglandin insert (Misodel®) have proved safe in American Studies and is registered in Denmark for use of induction. Misodel® was not included in RADS's evaluation, as there are only few studies on the effectiveness and side effects.

In the current study, investigators want to compare two different regimes for the induction of primipara who use respectively Misodel® and Angusta® as the primary method. The study is based on prospective collection of data from three divisions in Region Zealand, where investigators primarily compare the efficacy and safety but also to evaluate women's experience, the cost of medicine and consumption of resources in the maternity wards.

DETAILED DESCRIPTION:
Background The incidence of induced labour in Denmark, has increased from 12% in year 2000 to 25%, in 2014.

This increase is primarily due to a policy of earlier induction in women with prolonged pregnancy expected to decrease the risk of intrauterine fetal death. The national guidelines were changed in 2012.

Aim of the study To compare a regimen with use of 25 mcg peroral misoprostol (Angusta®) to 200 mcg vaginal insert Misoprostol (Misodel®) in a population of nullipara with unripened cervix. The regimens are compared in terms of technology (efficacy and safety), organisation, economy and patient-satisfaction.

Patients:

In the region of Zeeland, there are 6360 births annually, and among these 1636 (25%) births are induced. Among primipara there were 493 (29%) inductions in 2013. The number covers all induced births, i.e. medically, balloon-catheter, and amniotomy. In Holbæk Hospital (2013), 373 women were induced and among these 190 were primipara. In Næstved Hospital the number of inductions were 393 and 177 were primipara.

Regimes for induction:

There exist a number of different regimes for induction of labour. When the cervix is unripened, there is general consensus that the induction should be with either prostaglandins or a balloon catheter.

A committee appointed by Danish Regions (RADS) launched in 2014 a recommendation for the use of prostaglandins for induction of labour.

The recommendations are summarized in Table 1. The recommendations conclude that Angusta® should be the first line treatment for induction of labour with prostaglandins.

Table 1: Prostaglandins for induction of labour Prostaglandin Trade name Approved in Ministry of health RADS recommendations Misoprostol tablets, 25 mcg Angusta® Not approved Recommended: (2 h x 8) Dinoproston vaginal tablet or gel 3 mg Prostin® Minprostin® Approved Can be used: (6 h x 3) Misoprostol vaginal tablet 25 mcg Approved Can be used: (4 h x 4) Misoprostol tablets, 50 mcg Approved Can be used: (4 h x 4) Misoprostol insert 200 mcg Misodel® Approved Not recommended Dinoproston insert 10 mg Propess® Approved Not recommended

The quality of the evidence and strength of the recommendations are based on the evaluation method of GRADE (Grading of recommendations Assessment, Development and Evaluation).

The conclusions are primary based on a Cochrane analysis from June 2014.

Conclusions from this analysis were:

* Oral Misoprostol is more effective than placebo, and leads to a lower risk of caesarean delivery than dinoproston.
* Oral Misoprostol is equally effective when administered vaginally, but increases the risk of a low Apgar score and post-partum bleeding.

Recently, the conclusions of the Cochrane analysis has been debated. It has been argued that the evidence of effectiveness/equivalence is based on studies where oral misoprostol has been used in high dosages (>25 mcg), whereas the studies that concluded an increased risk of complications, used small dosages.

Misodel®:

Misoprostol insert 200 mcg (Misodel®) is registered in Europe for the induction of labour. The effect and safety is documented in studies from the US.

One randomized controlled study published in 2008, compared vaginal insert of 50 and 100 mcg misoprostol to vaginal insert of 10 mg Dinoproston. The two primary outcomes were the duration from administration to delivery, and the frequency of caesarean sections (CS). It was found that 100 mcg misoprostol and 10 mg dinoprostone had about the same duration from start of induction to delivery, whereas 50 mcg misoprostol showed a prolonged duration. The frequencies of CS were the same.

In 2011, the results from another RCT were published, comparing vaginal misoprostol insert of 100, 150 and 200 mcg. It was found that the 200 mcg group delivered within 25,8 hours for nulliparous, and 14 hours for multiparous women. The rate of CS was increased in this group, due to affected fetal heart-rate, although not significant. There were no differences in neonatal outcome. Tachysystoli (hyper-stimulation) was more frequent, but fewer needed to be stimulated with oxytocin (49%).

One RCT from 2013 compared 200 mcg slow release misoprostol to 10 mg Dinoproston insert. Their results showed a shorter duration to delivery (21,5 vs 32,8 hours), and the same frequency of CS.

RADS did not include Misodel® in their analysis since they found no RCTs that investigated the effect vs. side-effect in Misodel® compared with other regimes. The background for not recommending it, was that there seemed to be a high risk of tachysystoli with CTG changes - although based on different dosages.

The current trial:

This study is designed to compare 2 different regimens for induction of labour in nullipara with an unripened cervix by the use of a medical health technology assessment.

Patients:

Inclusion criteria: Primipara, immature cervix (Bishop score < 4), gestational age > 37+0 weeks with a singleton pregnancy without suspicion of fetal growth retardation (SGA defined as birth-weight deviation ≤-22%), and no history of prelabor rupture of membranes (PROM). No GDM.

Exclusion criteria: GA < 37+0 weeks, multipara, multiple pregnancy, placenta previa, suspicion of SGA, PROM, and GDM.

Methods The obstetric departments in the Region of Zeeland, have elaborated a clinical guideline for Angusta® that is expected to be fully implemented in the Hospitals of Roskilde, Næstved and Nykøbing Falster in June 2015. The guideline is based on the recommendations from RADS.

The department of Obstetrics in Holbæk has developed another guideline where Misodel® is used as first line treatment in a selected population. The women giving birth in Roskilde, Næstved and Holbæk are comparable on a number of parameters (BMI, distance to hospital, smoking, frequency of CS, cup-delivery etc.). This data is already available.

The project is based on a prospective collection of data for induced labour in Roskilde, Næstved and Holbæk. Investigators will also collect corresponding data for spontaneous delivery at term in the three different departments.

Primary outcomes:

* Frequency of caesarean section.
* Frequency of hyperstimulation, defined as tachysystoly with > 5 contractions in 10 minutes over a period of 30 minutes. Indeterminate or abnormal CTG. Scalp-pH < 7,20 or umbilical cord pH < 7,10.
* Frequency of delivery within 24 hours after induction.

Secondary outcomes:

* Time from induction to delivery
* Daytime delivery (8am-7pm)
* Number of hours with Syntocinon stimulation
* Use of ballon-catheter
* Epidural
* Numbers and durations of contact to labour ward
* Number of vaginal explorations under active labour
* Duration of CTG monitoring
* Fever
* Expenses for medication per induction (prostaglandins, syntocinon, balloon-catheter)
* Patient experience (evaluated based on questionnaire)
* Midwife experience (evaluated based on questionnaire)
* Breastfeeding (questionnaire 3 months after delivery)

Statistical analysis:

Outcome will be compared for the two departments with calculation of Odds Ratio (OR), with 95% confidence intervals (CI).

There will be adjusted for confounders such as BMI, maternity age, birth weight, gestational age, indication for induction by logistical regression analysis.

Datasource:

Approval from data protection authorities have been applied for. Besides the questionnaires, information will be available from electronic patient-charts, including MILOU (a program that stores CTG electronically).

Material size and strength-calculations for the primary outcomes:

Material size is determined with the Kelsey method with a significance level of 5% and power of 80%. For a more effective trial, we would like to set the ratio at 2:1 in control:Misodel® group.

* Caesarean section: A difference in 2% is estimated to be relevant (an expected difference of 20 to 22%). We need to include 4150 induced births in the Misodel® group and 8300 patients in the control group.
* Hyperstimulation: a difference in the frequency if tachysystoli in 15% is estimated to be relevant (40 to 55%). We need to include 126 and 252 patients in the Misodel® and control group.
* Birth within 24 hours: A difference of 15% is estimated to be relevant, where the results will be as above (40 to 55%): 126 and 252 patients per group.
* We are planning on including 140 induced women in the Misodel® group, and 280 in the control group. After the inclusion of 70 women, investigators will perform an interims-analysis. The investigators are not expecting to see any significant differences in CS.

Timeline:

The guideline for induction with Misodel® will be implemented in Holbæk in November 2015. The prospective collection of data is expected to be commenced in November 2015, and finished when the number of patients needed is reached (according to the sample size-calculations), presumably 1-2 years. Questionnaires for patient satisfactory will be elaborated and validated in May 2015.

Financing and conflicts of interests:

There will be no additional costs for medications or staff in the hospital of Holbæk. Funding for the study will be applied for from private and public funds, none is paid for by any pharmaceutical company.

Lone Krebs, Morten Lebech and Lisbeth Jønsson declare no conflicts of interest.

Data:

Data will be collected and stored by Axelina Eriksson (AE) at Holbæk Sygehus, department of Gynaecology and Obstetrics, in a locked office for interns at the department. Questionnaires will be locked in a drawer to which only AE has the key. Personal electronical data will only be accessed when AE is alone in the office, and the collection of information will be stored at AEs' personal login teamsite. A backup USB key will be stored in the same locked drawer, as the questionnaires. When data is processed in the office, it will be anonymized, and will only leave the office after anonymization. The project is scheduled to finish in 1/12-17 - all personal sensitive data will be destroyed afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Primipara, immature cervix (Bishop score < 4), gestational age > 37+0 weeks with a singleton pregnancy without suspicion of fetal growth retardation (SGA defined as birth-weight deviation ≤-22%), and no history of prelabor rupture of membranes (PROM). No GDM.

Exclusion Criteria:

* GA < 37+0 weeks, multipara, multiple pregnancy, placenta previa, suspicion of SGA, PROM, and GDM.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Nulliparous women to term with immature cervix
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of caesarean section | 1,5 year
  No of patients with caesarean section, will be registered for every patient, in their chart after birth, and assessed after 1,5 year.
Hyperstimulation | 1,5 year
  No of patients with hyperstimulation will be registered in the patient chart and assessed after 1,5 year.
  Defined as tachysystoly with > 5 contractions in 10 minutes over a period of 30 minutes. Indeterminate or abnormal CTG. Scalp-pH < 7,20 or umbilical cord pH < 7,10.
Delivery within 24 hours | 1,5 year
  Number of patients with delivery within 24 hours after induction, will be registered in the patient chart, and assessed after 1,5 year

SECONDARY OUTCOMES:
Timeline | 1,5 year
  Number of hours from induction to delivery, daytime delivery
Cost of primary induction method | 1,5 year
  Cost of medication (DKK for primary method of induction ie. Angusta and Misodel)
Experience | 1,5 year
  Patient and midwife - questionnaire based
Staff hours | 1,5 year
  Number of hours with midwife and number of hours admitted in hospital
Additional medications/treatments cost | 1,5 year
  Price in DKK for additional medications or treatments for induction ie. oxytocin and ballon catheter

CONTACTS AND LOCATIONS:
Locations (1):
- Gynækologisk obstetrisk afdeling, Holbæk, Denmark

REFERENCES:
- [Derived] Hansen KH, Eriksson A, Jeppesen S, Jeppegaard M, Krebs L. Women's experiences of induction of labour with misoprostol tablets compared with vaginal insert. Dan Med J. 2023 Jan 24;70(2):A04220232. PMID 36892220
- [Derived] Eriksson A, Jeppesen S, Krebs L. Induction of labour in nulliparous women- quick or slow: a cohort study comparing slow-release vaginal insert with low-dose misoprostol oral tablets. BMC Pregnancy Childbirth. 2020 Feb 7;20(1):79. doi: 10.1186/s12884-020-2770-0. PMID 32033600